CLINICAL TRIAL: NCT05048563
Title: Open Label Prospective Observational Registry of Thiola EC Therapy
Brief Title: Registry of Thiola EC Therapy
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 20-00331
Record Dates: First submitted 2021-09-13; First posted 2021-09-17 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cystinuria
MeSH Terms: conditions — Cystinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thiola EC represents several modifications of Thiola that promise better, more efficacious therapy of cystinuria. First, pill size has changed from 100 mg to 300 mg, meaning that typical pill burden will be reduced from, on average, 10 pills per day to 3-5 pills per day. This change will be welcomed by patients whose fluid intake and administration of potassium citrate are daily impositions. Second, the preparation is now enteric-coated, formulated to offer delayed release of active tiopronin. Lastly, Thiola EC can be taken with food which is an improvement to the inconvenient dosing regimen of Thiola, which can only be taken one hour before, or two hours after meals. These changes may affect compliance and side effect profiles compared to those of Thiola. In combination with potassium citrate or other alkali preparations, adverse GI effects are relatively common in actively-treated patients with cystinuria. It is possible that GI side effects may be reduced by Thiola EC.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Patients with cystinuria and a history of kidney stones
3. Taking Thiola EC
4. Willing and able to provide consent

Exclusion Criteria:

1. Unable to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cystinuria on Thiola EC.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Wisconsin Stone Quality Of Life (WiSQoL) Score | Baseline
  The WiSQoL questionnaire is designed to understand the quality of life of patients with a history of kidney stones. There are 7 main questions that each have sub-questions. The questions are answered on a scale from 1 (very true / always or almost always) to 5 (not at all true / not at all, never). The total range of questions is 28-140; the lower the score, the worse the quality of life.
Wisconsin Stone Quality Of Life (WiSQoL) Score | Month 6
  The WiSQoL questionnaire is designed to understand the quality of life of patients with a history of kidney stones. There are 7 main questions that each have sub-questions. The questions are answered on a scale from 1 (very true / always or almost always) to 5 (not at all true / not at all, never). The total range of questions is 28-140; the lower the score, the worse the quality of life.
Wisconsin Stone Quality Of Life (WiSQoL) Score | Month 12
  The WiSQoL questionnaire is designed to understand the quality of life of patients with a history of kidney stones. There are 7 main questions that each have sub-questions. The questions are answered on a scale from 1 (very true / always or almost always) to 5 (not at all true / not at all, never). The total range of questions is 28-140; the lower the score, the worse the quality of life.
Wisconsin Stone Quality Of Life (WiSQoL) Score | Month 18
  The WiSQoL questionnaire is designed to understand the quality of life of patients with a history of kidney stones. There are 7 main questions that each have sub-questions. The questions are answered on a scale from 1 (very true / always or almost always) to 5 (not at all true / not at all, never). The total range of questions is 28-140; the lower the score, the worse the quality of life.
Wisconsin Stone Quality Of Life (WiSQoL) Score | Month 24
  The WiSQoL questionnaire is designed to understand the quality of life of patients with a history of kidney stones. There are 7 main questions that each have sub-questions. The questions are answered on a scale from 1 (very true / always or almost always) to 5 (not at all true / not at all, never). The total range of questions is 28-140; the lower the score, the worse the quality of life.
Short Form-36 Health Survey (SF-36v2) Score | Baseline
  Scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status.
Short Form-36 Health Survey (SF-36v2) Score | Month 6
  Scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status.
Short Form-36 Health Survey (SF-36v2) Score | Month 12
  Scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status.
Short Form-36 Health Survey (SF-36v2) Score | Month 18
  Scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status.
Short Form-36 Health Survey (SF-36v2) Score | Month 24
  Scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status.

CONTACTS AND LOCATIONS:
Overall Officials: David Goldfarb, MD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - NYU Langone Health, New York, New York
  - Duke University, Durham, North Carolina
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data, researchers who provide a methodologically sound proposal, and investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose will have access to the data upon reasonable request. Requests should be directed to david.goldfarb@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.